CLINICAL TRIAL: NCT03820284
Title: Association Between Helicobacter Pylori and Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa osman taha, Principal investigator, Assiut University
Other Study IDs: L23457
Record Dates: First submitted 2019-01-19; First posted 2019-01-29 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Helicobacter Infections
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Group A inflammatory bowel disease with helicobacter pylori infection
- Group B: Inflammatory bowel disease without helicobacter pylori infection

SUMMARY:
Introduction:

Helicobacter pylori has been linked to a variety of gastric and extra gastric diseases. Chronic infection with H. pylori causes histologically evident gastritis in all colonized individuals and is the predominant risk factor for gastric and duodenal ulcers as well as gastric adenocarcinoma. However, increasingly robust experimental and epidemiological evidence suggests that H. pylori may at the same time be beneficial to its carriers, as it efficiently prevents allergic disorders and chronic inflammatory conditions .

Inflammatory bowel disease (IBD) is characterized by chronic, nonspecific intestinal inflammation with an unexplained pathology and an alternating relapsing and remitting clinical progression. IBD is divided into two subtypes: ulcerative colitis (UC) and Crohn's disease (CD). Most studies in the IBD field attribute its etiology to the complex interactions among immune dysfunction, genetic susceptibility of the host, and environmental risk factors.

Since the twenty-first century, improving hygienic conditions and socioeconomic status have reduced the H. pylori infection rate and this trend has concurrently been accompanied by an increased IBD incidence in most countries Numerous studies have reported a lower H. pylori infection rate in patients with CD and/or UC than in non-IBD control individuals. although a small number of studies showed no significant association .Recently, emerging epidemiologic studies and animal experiments revealed an inverse correlation between H. pylori infection and IBD onset, suggesting that H. pylori colonization exerts a special protective effect on autoimmune diseases

observation Cross sectional study will be conducted at assuit university hospitals on all patients with inflammatory disease to detect the prevalence of helicobacter pylori among them .Then the examined patients will be divided in to two group receiving the same medication group A : inflammatory bowel disease patient with H.PYLORI group B: inflammatory bowel disease Patient without H.PYLORI longitudinal study will be conducted to both group to study the clinical outcomes in both group .

DETAILED DESCRIPTION:
PATIENT AND METHOD :

observation Cross sectional study will be conducted at assuit university hospitals on all patients with inflammatory disease to detect the prevalence of helicobacter pylori among them .Then the examined patients will be divided in to two group receiving the same medication group A : inflammatory bowel disease patient with H.PYLORI group B: inflammatory bowel disease Patient without H.PYLORI longitudinal study will be conducted to both group to study the clinical outcomes in both group .

1. Thorough medical history and full clinical examination will be taken from all patient including

   -Personal history focus on special habit especially smoking

   -documented previous history for H.pylori eradication
   * Onset and duration of inflammatory bowel disease
   * current medication
   * presence of any extra intestinal manifestation of Inflammatory bowel disease
   * presence of any complications from Inflammatory bowel disease
2. Investigation :

   -All patients with inflammatory bowel disease will be tested for presence or absence of H.PYLORI by histological examination of endoscopically biopsied gastric mucosa

   -his to logical examination of colonic mucosal every 3 months

   -complete blood count

   -serum albumin

   -c reactive protein, erythrocyte sedimentation rate (ESR).

   -fecal calprotectin if possible
   * assess the severity of among both group (A,B) every 3 month for 2years. ulcerative by Mayo Score/Ulcerative Colitis Disease Activity Index and Crohn's disease by Montreal classifications for Crohn's Disease .

   Mayo Score/Ulcerative Colitis Disease Activity Stool frequency 0 = Normal 1 = 1-2 stools/day more than normal 2 = 3-4 stools/day more than normal 3 = 4 stools/day more than normal Rectal bleeding 0 = None 1 = Visible blood with stool less than half the time 2 = Visible blood with stool half of the time or more 3 = Passing blood alone Mucosal appearance at endoscopy 0 = Normal or inactive disease 1 = Mild disease (erythema, decreased vascular pattern, mild friability) 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions) 3 = Severe disease (spontaneous bleeding, ulceration) Physician rating of disease activity 0 = Normal 1 = Mild 2 = Moderate 3 = Severe

ELIGIBILITY:
Inclusion Criteria:

* all inflammatory bowel disease at assiut university will be included and examined in cross sectional study for detection of presence of H.pylori in one year 2019-2020 .then the examined patients will be divided in two group A ,B according to presence or absence of H pylori . Both group will be studied in cohort study for two years

Exclusion Criteria:

* -patients with history of administration of proton pump inhibitor or antibiotics with in eight weeks .
* patients with history of recent upper gastrointestinal bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inflammatory bowel disease patients with or without H.pylori infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
prevalance of H.pylori among patients with inflammatory bowel disease | One years
  Number of patient with inflammatory bowel disease with H.pylori infection
Mayo score activity index among ulcerative colitis patients with H.pylori and without H.pylori | Two years
  Stool frequency 0 = Normal 1 = 1-2 stools/day more than normal 2 = 3-4 stools/day more than normal 3 = 4 stools/day more than normal Rectal bleeding 0 = None 1 = Visible blood with stool less than half the time 2 = Visible blood with stool half of the time or more 3 = Passing blood alone Mucosal appearance at endoscopy 0 = Normal or inactive disease 1 = Mild disease (erythema, decreased vascular pattern, mild friability) 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions) 3 = Severe disease (spontaneous bleeding, ulceration) Physician rating of disease activity 0 = Normal 1 = Mild 2 = Moderate 3 = Severe
Mucosal healing among inflammatory bowel disease with H.pylori and without H.pylori | 1years
  Histological examination of the biopsied colonic mucosal every 3 months in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa Os Taha, Master of internal medicine, Principal Investigator — Assiut University; Zain elabdeen Ah Sayed, Doctorate of internal medicine, Study Director — Assiut; Alaa El Abdelmonem, Doctorate of internal medicine, Study Chair — Assiut University
Locations (1):
- Bahaa osman taha, Asyut, Egypt